CLINICAL TRIAL: NCT03723460
Title: Development of a Passive Dietary Monitoring System to Estimate an Individual's Dietary Intake in Households in Low and Middle-income Countries
Brief Title: Passive Dietary Intake Assessment Study
Acronym: PDIAS
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: KEMRI-Wellcome Trust Collaborative Research Program (Other); University of Ghana (Other); University of Pittsburgh (Other); Baylor College of Medicine (Other); University of Alabama at Birmingham (Other); Boston University (Other); University of Colorado, Denver (Other); University of Georgia (Other)
Responsible Party: Sponsor
Other Study IDs: 18IC4780; OPP1171395 (Other Grant/Funding Number: Bill & Melinda Gates Foundation)
Record Dates: First submitted 2018-10-25; First posted 2018-10-29 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Dietary Intake Assessment; Passive Dietary Monitoring; Malnutrition
Keywords: Dietary Intake Assessment; Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Households: Household here means a family unit comprising of at least both parents (mother and father) and a child under 5 years of age or an adolescent child.
  Interventions: Other: Passive Dietary Monitoring

INTERVENTIONS:
Other: Passive Dietary Monitoring — Passive dietary monitoring devices will be used to monitor dietary intake in household in communities in Ghana and Kenya

SUMMARY:
Currently, there is no accurate measurement of dietary intake. All current methodologies of assessing dietary intake have inaccuracy rates of 30 -70%. Accurate assessment of dietary intake is critical in understanding individual and population nutritional status and monitoring the effectiveness of public health interventions to maintain nutritional health. Estimating dietary intake in low and middle-income countries (LMICs) is remarkably challenging, albeit the high presence of malnutrition and the critical need for evidence-based data to inform policies and programmes on nutrition and health.

This study aims to develop and validate a low-cost and robust system for accurate measurement of an individual's dietary intake in households in LMICs. This innovative system passively recognises food, records intake, and estimates nutrient content of food. The system will be validated in field trials in Ghana and Kenya.

DETAILED DESCRIPTION:
This protocol describes the process of developing and validating a passive dietary monitoring system for the assessment of an individual's dietary intake in households in Ghana and Kenya.

The first phase of the study involves preliminary testing of identified dietary monitoring camera/video devices in a lab setting at Imperial College London under conditions similar to those anticipated in Ghana and Kenya. These conditions may include low lighting, unique foods common to certain regions, communal eating (where more than one person eats from a shared plate of cooked food) and placement of the devices on the body. This is important to guide the design of a suitable passive dietary monitoring system.

The second phase of the study involves an in-depth understanding of household set-up, composition and eating behaviour and testing the feasibility and acceptability of using passive dietary monitoring devices/system in communities in Ghana and Kenya. The data gathered in this phase of the study will inform the choice of the passive dietary monitoring system and configuration to use in the field validation study.

Finally, in the validation phase of the study, the passive dietary monitoring system developed will be set up to record food intake and estimate nutrient content of food across 88 households in Ghana and Kenya. In addition, 24h dietary recall (a commonly used method of collecting dietary intake data in population studies) and weighed food records will be used to estimate food intake in the households. The dietary intake data obtained through the passive monitoring system will be compared to 24h dietary recall and weighed food record data to validate its accuracy.

ELIGIBILITY:
Inclusion Criteria:

1. Household comprising of both parents (mother and father) and at least a child/children under 5 years of age and/or an adolescent child
2. Members of the household eat the same prepared meal
3. Willingness to use a camera/video recording device to capture household food preparation and consumption.

Exclusion Criteria:

* Households not meeting the above inclusion criteria will not be recruited

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population comprises of members of households living in rural and urban/per-urban communities in Ghana and Kenya
Sampling Method: Non-Probability Sample
Enrollment: 264 (Estimated)
Dates: Start 2018-11-15 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Dietary Intake Measures | 18 months
  This involves the use of camera/video imaging to estimate food volume/quantity, portion size (amount of ingested food) and nutrient content of food (macro and micronutrient content of food)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Frost, PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised individual participant data will be shared to other researchers through a secure cloud data storage system and through publication in open access journals.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 01 July 2020 - 30 January 2025
Access Criteria: Anonymised individual participant data will be shared to other researchers through a secure cloud data storage system and through publication in open access journals.

REFERENCES:
- [Derived] Jobarteh ML, McCrory MA, Lo B, Sun M, Sazonov E, Anderson AK, Jia W, Maitland K, Qiu J, Steiner-Asiedu M, Higgins JA, Baranowski T, Olupot-Olupot P, Frost G. Development and Validation of an Objective, Passive Dietary Assessment Method for Estimating Food and Nutrient Intake in Households in Low- and Middle-Income Countries: A Study Protocol. Curr Dev Nutr. 2020 Feb 7;4(2):nzaa020. doi: 10.1093/cdn/nzaa020. eCollection 2020 Feb. PMID 32099953